CLINICAL TRIAL: NCT05142969
Title: Effect of Chlorhexidine Bathing on Prevention of Hospital-Acquired Infections in Patients After Surgery in ICU: A Prospective, Single-Center, Single-Blind, Randomized Controlled Trial
Brief Title: Chlorhexidine Bathing to Prevent Hospital-acquired Infections: the CLEANS Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020ZSLC69
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Chlorhexidine; Hospital-Acquired Infection; Surgery; Intensive Care Unit
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients were daily bathed with soap and water only.
- Intervention arm (Experimental): Patients were daily bathed with soap and water and then receive 2% Chlorhexidine bathing (Petel Skin care wipes, Likang LtD, shanghai, China).
  Interventions: Other: 2% Chlorhexidine bathing

INTERVENTIONS:
Other: 2% Chlorhexidine bathing — Eight chlorhexidine-impregnated cloths are used in sequential order to wipe the body surfaces from neck to toe to avoid exposure of chlorhexidine to the mucous membranes of the eyes, ears and mouth.
  Arms: Intervention arm

SUMMARY:
Hospital-acquired infections (HAI) have been shown to increase length of hospital stay and mortality. Infections acquired during a hospital stay have been shown to be preventable. The skin of patients is considered a major reservoir for pathogens associated with hospital-acquired infections, and has been suggested as a potential target for interventions to reduce bacterial burden and subsequent risk of infection. The use of daily Chlorhexidine (CHG) bathing in intensive care patients has been advocated to reduce many of the infections in critically ill patients. However, the effectiveness of CHG bathing to reduce ICU infections has varied considerably among published trials, making the effectiveness of CHG bathing in ICU patients uncertain.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥ 18-years old)
* anticipated SICU stay for 48 hours or more
* APACHE II >15

Exclusion Criteria:

* Braden Scale for Predicting Pressure Sore Risk score more than 9 (highest risk)
* pregnancy
* skin irritation
* chlorhexidine allergy
* SICU stay of more than 48 hours prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital-acquired infections | throughout study completion, an average of 7 days
  Including bloodstream infections (BSI), central line-associated BSI (CLABSI), ventilator-associated pneumonia (VAP) and catheter-associated urinary tract infection (CAUTI).

SECONDARY OUTCOMES:
Multidrug-resistant bacterial colonization free time | throughout study completion, an average of 7 days
  Time that the swab samples collected from axilla and groin were persistently negative for target MDR throughout ICU admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China